CLINICAL TRIAL: NCT06240715
Title: A Cluster Randomized Clinical Trial of Umbilical Cord Milking Compared to Early Cord Clamping in Preterm Infants Who Are Non-vigorous at Birth
Brief Title: Comparative Outcomes Related to Delivery-room Cord Milking In Low-resourced Kountries- PreTerm
Acronym: CORDMILK-PT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Thrasher Research Fund (Other); Thomas Jefferson University (Other); Sharp HealthCare (Other); Jawaharlal Nehru Medical College (Other); Daga Memorial Maternity and Children's Hospital, Nagpur, India (Unknown); Mahatma Gandhi Institute of Medical Sciences, Wardha, India (Unknown); Indira Gandhi Government Medical College & Hospital, Nagpur, India (Unknown); Pimpri Chinchwad Municipal Corporation's Post-Graduate Institute, Yashwantrao Chavan Memorial Hospital, Pune, India (Unknown); Government Medical College, Nagpur (Industry); Government Medical College, Chandrapur, India (Unknown); Osmania Medical College, Niloufer Hospital, Hyderabad, India (Unknown)
Responsible Party: Principal Investigator, Zubair Aghai, Professor of Pediatrics, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CORDMILK-PT
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Preterm; Infant Death
Keywords: Preterm; Umbilical cord milking; Placental transfusion
MeSH Terms: conditions — Premature Birth; Infant Death; Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Crossover
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Active Comparator): The delivering practitioner will place the newborn below the level of the incision (at the edge of the table) at C/S and a second team member will milk the cord four times. For vaginal delivery, the delivering obstetrician, midwife or perinatal provider will hold the infant against their body or place the infant on the mother's abdomen and the cord will be milked either four times by the obstetrical provider or by a second team member. For the cord milking procedure, the obstetrical provider will milk 20-30 centimeters length of the umbilical cord over two seconds, repeating three additional times as described previously. This time is not significantly different from the time for early cord clamping (ECC).
  Interventions: Procedure: Umbilical cord milking
- Early Cord Clamping (No Intervention): Umbilical cord will be clamped immediately after birth (within 60 seconds)

INTERVENTIONS:
Procedure: Umbilical cord milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 1--15 seconds.
  Other Names: UCM
  Arms: Umbilical Cord Milking

SUMMARY:
The goal of this multicenter, cluster-randomized, crossover trial is to determine if umbilical cord milking compared to early cord clamping will reduce in-hospital mortality in non-vigorous preterm infants born between 30 weeks and 34 weeks of gestation.

DETAILED DESCRIPTION:
Background: Prematurity is the leading cause of death in children younger than 5 years of age. Worldwide, 15 million infants are born premature, and India alone contributes to quarter of them. Approximately 1 million children die each year due to complications of prematurity.

Delayed cord clamping (DCC), one of the methods of transfer of placental blood to neonates (placental transfusion) immediately after birth reduce mortality by 30% in premature infants. But DCC is not recommended in neonates who require immediate resuscitation. Umbilical cord milking (UCM) is an option for placental transfusion in preterm infants who require immediate resuscitation but not currently recommended due to lack of randomized clinical trials.

HYPOTHESIS: UCM will reduce the in-hospital mortality in non-vigorous preterm infants born between 30 weeks to 34 weeks of gestation compared to early cord clamping.

METHODS: This multicenter cluster crossover randomized trial will enroll approximately 800 preterm infants to early cord clamping or milking the intact cord 4 times prior to clamping.

IMPACT: If investigators find that UCM is beneficial, this simple, low-tech, no cost intervention can be used in preventing deaths in preterm infants. This trial will potentially provide evidence to support a change in guidelines making UCM part of standard practice worldwide for preterm infants who require immediate resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 30 0/7 weeks to 34 6/7 weeks of gestation
* Non-vigorous at birth

Exclusion Criteria:

* Infants with congenital malformation
* Major chromosomal abnormalities
* Complete placental abruption/cutting through the placenta at the time of delivery
* Cord conditions (umbilical knots, inadequate cord length, cord rupture, non-reducible nuchal cord)
* Mono-chorionic twins,
* Twins with no information on amnion/chorion
* Multiple gestation >2

Ages: 0 Minutes to 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | From date of birth until the date of discharge from the hospital or date of death from any cause, whichever come first, assessed up to 12 weeks
  Death of a baby during birth hospitalization

SECONDARY OUTCOMES:
Hemoglobin at or after 24 hours | Days 1-7
  Hb levels
Early and late onset culture positive sepsis | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of infants with early onset or late onset sepsis
Any intraventricular hemorrhage (IVH) and severe IVH (grade 3 or 4) | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of infants with any IVH or severe IVH
Need for blood transfusion | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of infants received blood transfusion
Moderate to severe hypoxemic ischemic encephalopathy | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of infants with moderate to severe hypoxemic ischemic encephalopathy
Necrotizing enterocolitis (Bell's stage 2 or higher) | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of infants with necrotizing enterocolitis (Bell's stage 2 or higher)
Need for medications for hypotension | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of infants needed medications for hypotension
Need for phototherapy for jaundice | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of infants needed phototherapy for jaundice
Retinopathy of prematurity (ROP) requiring intervention | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of infants with ROP that required intervention
Length of hospitalization | From date of birth until the date of discharge from the hospital, assessed up to 12 weeks.
  Number of days infants stayed in hospital

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - KLE Academy of Higher Education and Research (Deemed-to-be-University) Jawaharlal Nehru Medical College, Belagavi, Karnataka
  - Government Medical College, Chandrapur, Maharashtra
  - Indira Gandhi Government Medical College & Hospital, Nagpur, Maharashtra
  - Yashwantrao Chavan Memorial Hospital, Pune, Maharashtra
  - Daga Memorial Woman and Children Hospital, Nagpur, MS
  - Government Medical College and Hospital, Nagpur, MS
  - Mahatma Gandhi Institute of Medical Sciences/ Kasturba Hospital, Wardha, MS
  - Sawai Man Singh Medical College, Jaipur, Rajasthan
  - Osmania Medical College, Niloufer Hospital, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: Yes